CLINICAL TRIAL: NCT03230734
Title: Randomized, Multicentre Phase II Trial of the Sequencing of Radium-223 and Docetaxel Plus Prednisone in Symptomatic Bone-only Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Sequencing of Radium-223 and Docetaxel in Symptomatic Bone-only Metastatic Castration-resistant Prostate Cancer
Acronym: RAPSON
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRST185.04; 2016-004452-29 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: prostate cancer; castration-resistant prostate cancer; metastatic prostate cancer; bone only metastatic prostate cancer; radium-223; Docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm A (Experimental): radium-223 initially followed by docetaxel plus prednisone at the time of progression (PD)
  Interventions: Drug: Radium-223; Drug: Docetaxel
- Treatment Arm B (Experimental): docetaxel plus prednisone initially followed by radium-223 at the time of progression (PD)
  Interventions: Drug: Radium-223; Drug: Docetaxel

INTERVENTIONS:
Drug: Radium-223 — Radium-223: administered at the dose of 55 kBq per kg body weight, given at 4 week intervals for 6 injections, by slow intravenous injection
Drug: Docetaxel — Docetaxel: administered at the dose of 75 mg/m2 by intravenous infusion over a period of 1 hour every 3 weeks for 10 cycles. It is associated with prednisone 5 mg orally twice daily administered continuously.

SUMMARY:
Randomized, multicentre phase II trial of the sequencing of Radium-223 and Docetaxel plus prednisone in symptomatic bone-only metastatic castration-resistant prostate cancer (mCRPC)

Open-label, randomized phase II trial in patients with symptomatic bone-only metastatic castration-resistant prostate cancer. Eligible patients are randomly assigned into two arms:

* Arm A: radium-223 initially followed by docetaxel plus prednisone at the time of progression (the second step is optional according to clinical evolution of disease)
* Arm B: docetaxel plus prednisone initially followed by radium-223 at the time of progression (the second step is optional according to clinical evolution of disease).

DETAILED DESCRIPTION:
Randomized, multicentre phase II trial of the sequencing of Radium-223 and Docetaxel plus prednisone in symptomatic bone-only metastatic castration-resistant prostate cancer (mCRPC) Primary objective: To determine the effects of sequential treatment between radium-223 and docetaxel on the percentage of symptomatic bone-only CRPC patients experiencing improvement or worsening in health-related quality of life (HRQoL) Secondary objective: To compare survival in patients treated with sequential therapy between radium-223 and docetaxel and to identify predictive factors of Radium-223 for clinical outcome (progression free survival and overall survival) in this patient population.

Study Treatment:

Radium-223: administered at the dose of 55 kBq per kg body weight, given at 4 week intervals for 6 injections, by slow intravenous injection.

Docetaxel: administered at the dose of 75 mg/m2 by intravenous infusion over a period of 1 hour every 3 weeks for 10 cycles. It is associated with prednisone 5 mg orally twice daily administered continuously.

Statistical methodology A responder analysis investigating treatment effects on percentage of patients experiencing meaningful HRQoL improvement/worsening on treatment will be conducted. When defining meaningful improvement/worsening, the upper limit of the minimally important difference (MID) range will be used. The MIDs for FACT-P total score and subscales that will be used in this study will be 10 and 3, respectively.

Patients experiencing a QoL increase >=MID from baseline at week 12 will be considered responders while patients experiencing a decrease in HRQoL score >=MID at this time point will be considered to have experienced worsening HRQoL.

According to primary endpoint, considering a type I error 0.10, type II error 0.20, proportion of responder patients in the standard arm 0.10 and in the experimental arm of 0.40, a total of 70 patients (35 for each arm) will be enrolled in the study. Chi-square tests will be used to test for an association between treatment and meaningful improvement (i.e. responder) or worsening in HRQoL.

According to secondary endpoints, PFS, TPFS and OS will be estimated by the Kaplan-Meier method. The treatment groups will be compared with a two-sided log rank test. All analyses will be done in the intention-to-treat population. For translational studies, we will conduct a prognostic and predictive factor analysis for time-to-event clinical outcomes using a univariate Cox model; significant factors subsequently will be included in a multivariable Cox regression model (cutoff p<0•05).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed adenocarcinoma of prostate
2. Two or more bone metastases confirmed by bone scintigraphy within 8 weeks prior to randomization
3. Symptomatic disease defined as regular use of opioid or nonopioid analgesic medication or treatment with external beam radiation therapy within the previous 12 weeks for cancer-related bone pain
4. Known castration-resistant disease, defined according to PCWG3 criteria (59) as: castrate serum testosterone level: ≤50 ng/dL (≤1.7 nmol/L)
5. Subjects who have failed initial hormonal therapy, either by orchiectomy or by using a GnRH agonist in combination with an anti-androgen, must first progress through antiandrogen withdrawal prior to being eligible. The minimum timeframe to document failure of anti-androgen withdrawal will be four weeks
6. Progressive disease based on PSA and/or radiographic PCWG3 criteria:

   a. Serum PSA progression defined as two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least one week apart. Serum PSA at screening ≥ 1ng/mL is the minimal starting value b. or radiographic disease progression based on documented bone lesions by the appearance of two or more new lesions by bone scintigraphy.
7. Patients who failed treatment with any ADT, abiraterone and/or enzalutamide for CRPC that must be terminated at least 4 weeks beforeC1D1.
8. Patients who received prior docetaxel for hormone-naïve prostate cancer should only be allowed if more than 2 years have been between the last administration of docetaxel and C1D1.
9. Male, aged ≥18 years
10. Life expectancy of greater than 6 months
11. ECOG performance status≤2 (see Appendix A)
12. Patients must have normal organ and marrow function as defined below:

    * leukocytes > 3,000/µL
    * absolute neutrophil count >1,500/µL
    * platelets >100,000/µL
    * total bilirubin within normal institutional limits
    * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
    * creatinine within normal institutional limits In the presence of borderline values, the participating Centers will be able to discuss individual cases with the Coordinating Center.
13. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after the last dose of radium-223 or docetaxel, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (2020_09) (See Appendix F). Two acceptable methods of birth control thus include condom (barrier method of contraception) and one of the following is required (established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy), for more than 6 months.
14. No evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).
15. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Patients who have had radiotherapy within 4 weeks prior to C1D1.
2. Patients with known visceral metastases
3. Participation in another clinical trial with any investigational agents within 30 days prior to C1D1.
4. Concurrent use of other anticancer agents or treatments, with the following exceptions: LHRH agonists or antagonists, denosumab or bisphosphonate (eg, zoledronic acid). Ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients who received systemic radiotherapy (e.g. samarium, strontium etc.) for the treatment of bone metastases.
7. Patients who received blood transfusion or erythropoietin within the last 4 weeks prior to start of study treatment.
8. Patients who received prior treatment with Radium-223.
9. Patients with malignant lymphadenopathy exceeding 3 cm in short-axis diameter, or symptomatic nodal disease, i.e. scrotal, penile or leg edema.
10. Other primary tumor (other than CRPC) including hematological malignancy present within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer).
11. Maintenance treatment with corticosteroids corresponding to a prednisolone or prednisone dose above 10 mg/day. The dose must have been stable for at least 5 days.
12. Patients with imminent or established spinal cord compression based on clinical findings and/or magnetic resonance imaging.
13. Positive test for HIV in case of known positivity to human immunodeficiency virus (HIV).

    * Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen[HBsAg] test at screening) or hepatitis C Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life (HRQoL) clinical benefit | up to 36 months
  HRQoL clinical benefit, according to the Functional Assessment of Cancer Therapy-Prostate (FACT-P)
health-related quality of life (HRQoL ) clinical benefit | up to 36 months
  HRQoL clinical benefit, according to Brief Pain Inventory-Short Form questionnaire (BPI) for bone pain intensity.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 36 months
  PFS defined as the duration of time from randomization to time of progression or death, whichever occurred earlier
Total progression-free survival (TPFS) | up to 36 months
  TPFS defined as total PFS at the end of the therapeutic sequence
Overall survival (OS) | up to 36 months
  OS defined as the time from randomization to the date of death due to any cause or the last date the patient was known to be alive
toxic effects categorization for safety monitoring | up to 36 months
  evaluation of toxicity by Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Identification of markers predictive to clinical outcome | up to 36 months
  Identification of markers predictive to clinical outcome including:
  * translational studies of circulating tumor DNA and/or circulating tumor cells and/or circulating RNA
  * serum chromogranin A and neuron specific enolase levels
  * positron emission tomography (PET) with choline and/or new tracer

CONTACTS AND LOCATIONS:
Overall Officials: Ugo De Giorgi, MD, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Via Maroncelli 40, 47014 Meldola, ITALY
Locations (15):
- Italy (15):
  - UO Oncologia Medica, IRST IRCCS, Meldola, FC
  - U.O. Oncologia PO Vito Fazzi, Lecce, LE
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - UO Oncologia Medica, C.R.O.B. - I.R.C.C.S, Rionero in Vulture, PZ
  - Ospedale S. Chiara - UO Oncologia Medica, Trento, TN
  - Oncologia Medica San Luigi Gonzaga, Orbassano, TO
  - Ospedale Sacro Cuore "Don Calabria", Negrar, VR
  - UO Oncologia medica, IRCCS Centro di Riferimento Oncologico di Aviano, Aviano
  - IO Oncologia Medica, Ospedale Regionale Bolzano - Az. Sanitaria Alto Adige, Bolzano
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Istituto Europeo di Oncologia, Milan
  - INT di Napoli Fondazione "G. Pascale", Napoli
  - UO Oncologia Medica, Azienda Ospedaliera-Universitaria di Parma, Parma
  - UO Oncologia Medica, AOU PISANA - Ospedale Santa Chiara, Pisa
  - Azienda Ospedaliera Arcispedale S. Maria Nuova/IRCCA di Reggio Emilia, Reggio Emilia